CLINICAL TRIAL: NCT01737697
Title: Multicenter, Two-phase, Multi-dose, Prospective, Randomized, Double-blind, Placebo-Controlled Study of Safety and Efficacy of Microporous, Fractionated, Protonated Zirconium Silicate in Mild to Moderate Hyperkalemia
Brief Title: Safety & Efficacy of Zirconium Silicate in Mild to Moderate Hyperkalemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZS Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ZS-003
Record Dates: First submitted 2012-11-19; First posted 2012-11-29 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Hyperkalemia
MeSH Terms: conditions — Hyperkalemia | interventions — zircon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Zirconium silicate (acute phase) (Experimental): Randomized oral doses (1.25g, 2.5g, 5g, and 10g) of microporous, fractionated, protonated zirconium silicate administered 3 times (tid) daily with meals for 48 hours.
  Interventions: Drug: Zirconium silicate (acute phase)
- Placebo (acute phase) (Placebo Comparator): Placebo ( silicified microcrystalline cellulose) randomized to mimic doses of experimental drug administered 3 times (tid) daily with meals.
  Interventions: Drug: Placebo (acute phase)
- Zirconium silicate (subacute phase) (Experimental): Randomized oral doses (1.25g, 2.5g, 5g, and 10g) of microporous, fractionated, protonated zirconium silicate administered once a day prior to the morning meal for 12 days.
  Interventions: Drug: Zirconium silicate (subacute phase)
- Placebo (subacute phase) (Placebo Comparator): Placebo (silicified microcrystalline cellulose) randomized to mimic doses of experimental drug administered once a day (qd) prior to the morning meal for 12 days.
  Interventions: Drug: Placebo ( subacute phase)

INTERVENTIONS:
Drug: Zirconium silicate (acute phase) — Randomized oral doses (1.25g, 2.5g, 5g, and 10g) of microporous, fractionated, protonated zirconium silicate administered 3 times (tid) daily with meals for 48 hours.
  Other Names: ZS
  Arms: Zirconium silicate (acute phase)
Drug: Zirconium silicate (subacute phase) — Randomized oral doses (1.25g, 2.5g, 5g, and 10g) of microporous, fractionated, protonated zirconium silicate administered once a day prior to the morning meal for 12 days.
  Other Names: ZS
  Arms: Zirconium silicate (subacute phase)
Drug: Placebo (acute phase) — Randomized to mimic doses of experimental drug administered 3 times (tid) daily with meals for 48 hours during the acute phase.
  Other Names: Silicified microcrystalline cellulose
  Arms: Placebo (acute phase)
Drug: Placebo ( subacute phase) — Randomized to mimic doses of experimental drug administered once a day prior to the morning meal for 12 days during the subacute phase.
  Other Names: Silicified microcrystalline cellulose
  Arms: Placebo (subacute phase)

SUMMARY:
Acute Phase: It is hypothesized that ZS (zirconium silicate) is more effective than placebo control (alternative hypothesis) in lowering S-K levels in subjects with S-K between 5.0 - 6.5 mmol/l versus no difference between ZS and placebo control (null hypothesis).

Subacute Phase (randomized withdrawal): It is hypothesized that ZS once daily is more effective than placebo control (alternative hypotheses) in maintaining normokalemic levels (3.5 - 4.9 mmol/l) among subjects completing the Acute Phase versus no difference between each ZS dose and respective placebo controls (null hypotheses).

DETAILED DESCRIPTION:
A total of 750 subjects with mild to moderate hyperkalemia (i- STAT potassium levels between 5.0-6.5 mmol/l, inclusive) will be enrolled in the study where they, in a double-blind fashion, will be randomized 1:1:1:1:1 to receive one of four (4) doses of ZS (1.25g, 2.5g, 5g, and 10g) or placebo control, administered 3 times daily (tid) with meals for the initial 48 hours (Acute Phase), followed by a Subacute Phase (randomized withdrawal) during which patients treated with active doses in the Acute Phase, who achieve normokalemia (i-STAT potassium values 3.5 to 4.9 mmol/l, inclusive) will be randomized to 12 days of subacute, once a day (qd) dosing. There will be a one-time randomization to assign the Acute Phase treatment and the Subacute Phase treatment. The Subacute Phase will include subjects who became normokalemic on active drug and those who became normokalemic on placebo. The former will be randomized in a 1:1 ratio between the same dose of ZS they received during the acute phase but only administered once a day (qd) or placebo, qd. Subjects on placebo during the Acute Phase who are normokalemic in the morning of Study Day 3, will be randomized to receive either 1.25 or 2.5 g ZS, qd as Subacute Phase treatment.

Safety and tolerability will be assessed on an ongoing basis by an Independent Data Safety Monitoring Board (DSMB). Each active dose group will consist of 150 patients per treatment group including the placebo control group for a total of 750 patients; the 1:1:1:1:1 allocation helps to optimize the multiple active dose comparisons to the respective placebo controls for the Subacute Phase.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent.
* Over 18 years of age.
* Mean i-STAT potassium values between 5.0 - 6.5 mmol/l inclusive, at screening (Study Day 0).
* Ability to have repeated blood draws or effective venous catheterization.
* Women of childbearing potential must be practicing a highly effective method of birth control.

Exclusion Criteria:

* Pseudohyperkalemia signs and symptoms, such as excessive fist clinching hemolyzed blood specimen, severe leukocytosis or thrombocytosis.
* Subjects treated with lactulose, xifaxan or other nonabsorbed antibiotics for hyperammonemia within the last 7 days.
* Subjects treated with resins (such as Sevelamer acetate or Sodium polystyrene sulfonate [SPS; e.g. Kayexalate®]), calcium acetate, calcium carbonate, or lanthanum carbonate, within the last 7 days.
* Subjects with a life expectancy of less than 3 months.
* Subjects who are HIV positive.
* Subjects who are severely physically or mentally incapacitated and who in the opinion of investigator are unable to perform the subjects' tasks associated with the protocol.
* Women who are pregnant, lactating, or planning to become pregnant.
* Subjects with Ketoacidosis/Acidemia.
* Presence of any condition which, in the opinion of the investigator, places the subject at undue risk or potentially jeopardizes the quality of the data to be generated.
* Known hypersensitivity or previous anaphylaxis to ZS or to components thereof.
* Previous treatment with ZS
* Treatment with a drug or device within the last 30 days that has not received regulatory approval at the time of study entry.
* Subjects with cardiac arrhythmias that require immediate treatment.
* Insulin-dependent diabetes mellitus
* Subjects on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 754 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2013-10-31 (Actual); Study Completion 2013-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Rasmussen, MD, Study Chair — ZS Pharma, Inc.
Locations (44):
- United States (42):
  - Pinnacle Research Group, Anniston, Alabama
  - Saadat Ansari Internal Medicine, Huntsville, Alabama
  - Aspire Clinical Studies, LLC, Glendale, Arizona
  - Southwest Clinical Research Institute, Tempe, Arizona
  - California Institute of Renal Research, Chula Vista, California
  - Torrance Clinical Research, Lomita, California
  - Academic Medical Research Institute, Los Angeles, California
  - Mohammad Ismail, Inc, Paramount, California
  - Apex Research of Riverside, Riverside, California
  - Capital Nephrology Clinical Group, Sacramento, California
  - Pikes Peak Nephrology Associates, Colorado Springs, Colorado
  - Denver Nephrologists, PC, Denver, Colorado
  - Nephrology and Hypertension Associates, Middlebury, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - Clinical Research of Brandon, Brandon, Florida
  - Meridien Research, Brooksville, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Endocrinology of Central Florida, Lake Mary, Florida
  - Meridien Research, Lakeland, Florida
  - San Marcus Research Clinic, Miami, Florida
  - Medical Consulting Center, Miami, Florida
  - Elite Research Institute, Miami, Florida
  - Prevention & Strengthening Solutions, Inc, Miramar, Florida
  - PCCC of Volusia, New Smyrna Beach, Florida
  - Meridien Research, St. Petersburg, Florida
  - Lakeview Medical Research, Summerfield, Florida
  - Clinical Research Trials of Florida, Tampa, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Research by Design, Evergreen Park, Illinois
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Washington Nephrology Associates, Bethesda, Maryland
  - Nephrology Center DBA, Paragon Health PC, Kalamazoo, Michigan
  - The Center for Clinical Trials, Biloxi, Mississippi
  - Clinical Research Consultants, LLC, Kansas City, Missouri
  - United Medical Associates, Binghamton, New York
  - Life Medi-Research and Management, Brooklyn, New York
  - Doylestown Hospital Medical Research, Doylestown, Pennsylvania
  - South Carolina Nephrology & Hypertension, Orangeburg, South Carolina
  - Carolina Diabetes and Kidney Center, Sumter, South Carolina
  - Southwest Houston Research, Ltd, Houston, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - Southern Utah Kidney and Hypertension Center, St. George, Utah
- Australia (2):
  - Renal Research, Gosford, New South Wales
  - Melbourne Renal Research Group, Reservoir, Victoria

REFERENCES:
- [Derived] Natale P, Palmer SC, Ruospo M, Saglimbene VM, Strippoli GF. Potassium binders for chronic hyperkalaemia in people with chronic kidney disease. Cochrane Database Syst Rev. 2020 Jun 26;6(6):CD013165. doi: 10.1002/14651858.CD013165.pub2. PMID 32588430
- [Derived] Amin AN, Menoyo J, Singh B, Kim CS. Efficacy and safety of sodium zirconium cyclosilicate in patients with baseline serum potassium level >/= 5.5 mmol/L: pooled analysis from two phase 3 trials. BMC Nephrol. 2019 Dec 2;20(1):440. doi: 10.1186/s12882-019-1611-8. PMID 31791288
- [Derived] Friedman PA, Scott CG, Bailey K, Baumann NA, Albert D, Attia ZI, Ladewig DJ, Yasin O, Dillon JJ, Singh B. Errors of Classification With Potassium Blood Testing: The Variability and Repeatability of Critical Clinical Tests. Mayo Clin Proc. 2018 May;93(5):566-572. doi: 10.1016/j.mayocp.2018.03.013. PMID 29728199
- [Derived] Packham DK, Rasmussen HS, Lavin PT, El-Shahawy MA, Roger SD, Block G, Qunibi W, Pergola P, Singh B. Sodium zirconium cyclosilicate in hyperkalemia. N Engl J Med. 2015 Jan 15;372(3):222-31. doi: 10.1056/NEJMoa1411487. Epub 2014 Nov 21. PMID 25415807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 65 sites (up to 100 sites initially planned in Protocol) in the United States, Australia, and South Africa from 25 November 2012 to 29 October 2013.
Pre-assignment Details: In the acute phase, 754 subjects were randomized; 753 were treated. Subjects who completed the AP and had i-STAT K+ values within normal range in a.m. of Study Day 3 could enter the Subacute Phase. 543 subjects entered the subacute phase.
Groups:
- Acute Phase: Placebo: Participants administered placebo as suspension orally three times a day (TID) for first 48 hours.
- Acute Phase: Sodium Zirconium Cyclosilicate (ZS) 1.25 g TID: Participants administered ZS 1.25 g TID as suspension orally for first 48 hours.
- Acute Phase: ZS 2.5 g TID: Participants administered ZS 2.5 g TID as suspension orally for first 48 hours.
- Acute Phase: ZS 5 g TID: Participants administered ZS 5 g TID as suspension orally for first 48 hours.
- Acute Phase: ZS 10 TID: Participants administered ZS 10 g TID as suspension orally for first 48 hours.
- Subacute Phase: Placebo Matched to ZS 1.25g QD: Participants who received ZS 1.25 g TID in the acute phase and administered placebo as suspension once daily (QD) for 12 days.
- Subacute Phase: ZS 1.25 g QD: Participants who received ZS 1.25g TID in the acute phase and administered ZS 1.25 g QD for 12 days.
- Subacute Phase: Placebo Matched to ZS 2.5 g QD: Participants who received ZS 2.5 g TID in the acute phase and administered placebo as suspension QD for 12 days.
- Subacute Phase: ZS 2.5 g QD: Participants who received ZS 2.5 g TID in the acute phase and administered ZS 2.5 g as suspension QD for 12 days.
- Subacute Phase: Placebo Matched to ZS 5 g QD: Participants who received ZS 5 g TID in the acute phase and administered placebo as suspension QD for 12 days.
- Subacute Phase: ZS 5 g QD: Participants who received ZS 5 g TID in the acute phase and administered ZS 5 g as suspension QD for 12 days.
- Subacute Phase: Placebo Matched to ZS 10 g QD: Participants who received ZS 10 g TID in the acute phase and administered placebo as suspension QD for 12 days.
- Subacute Phase: ZS 10 g QD: Participants who received ZS 10 g TID in the acute phase and administered ZS 10 g QD as suspension for 12 days.
- Subacute Phase: ZS 1.25 (Acute Phase: Placebo): Participants who received placebo in the acute phase and administered ZS 1.25 g as suspension QD for 12 days.
- Subacute Phase: ZS 2.5 g (Acute Phase: Placebo): Participants who received placebo in the acute phase and administered ZS 2.5 g as suspension QD for 12 days.
Period: Acute Phase-Initial 48 Hours
Arm/Group | Acute Phase: Placebo | Acute Phase: Sodium Zirconium Cyclosilicate (ZS) 1.25 g TID | Acute Phase: ZS 2.5 g TID | Acute Phase: ZS 5 g TID | Acute Phase: ZS 10 TID | Subacute Phase: Placebo Matched to ZS 1.25g QD | Subacute Phase: ZS 1.25 g QD | Subacute Phase: Placebo Matched to ZS 2.5 g QD | Subacute Phase: ZS 2.5 g QD | Subacute Phase: Placebo Matched to ZS 5 g QD | Subacute Phase: ZS 5 g QD | Subacute Phase: Placebo Matched to ZS 10 g QD | Subacute Phase: ZS 10 g QD | Subacute Phase: ZS 1.25 (Acute Phase: Placebo) | Subacute Phase: ZS 2.5 g (Acute Phase: Placebo)
Started | 158 | 154 | 141 | 158 | 143 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 157 | 150 | 137 | 152 | 140 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 4 | 4 | 6 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — hypo-or hyperkalemia | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Family emergency | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor's decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Subacute Phase
Arm/Group | Acute Phase: Placebo | Acute Phase: Sodium Zirconium Cyclosilicate (ZS) 1.25 g TID | Acute Phase: ZS 2.5 g TID | Acute Phase: ZS 5 g TID | Acute Phase: ZS 10 TID | Subacute Phase: Placebo Matched to ZS 1.25g QD | Subacute Phase: ZS 1.25 g QD | Subacute Phase: Placebo Matched to ZS 2.5 g QD | Subacute Phase: ZS 2.5 g QD | Subacute Phase: Placebo Matched to ZS 5 g QD | Subacute Phase: ZS 5 g QD | Subacute Phase: Placebo Matched to ZS 10 g QD | Subacute Phase: ZS 10 g QD | Subacute Phase: ZS 1.25 (Acute Phase: Placebo) | Subacute Phase: ZS 2.5 g (Acute Phase: Placebo)
Started | 0 | 0 | 0 | 0 | 0 | 41 | 49 | 46 | 54 | 68 | 65 | 61 | 63 | 46 | 50
Completed | 0 | 0 | 0 | 0 | 0 | 38 | 48 | 43 | 52 | 66 | 59 | 58 | 61 | 44 | 49
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 2 | 2 | 6 | 3 | 2 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 4 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Hypo-or hyperkalemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One subject in ZS 5g group was randomized but was not treated and is excluded from baseline characatertics.
Groups:
- Acute Phase: Placebo TID: Participants administered placebo three times daily (TID) orally as suspension for first 48 hours.
- Total: Total of all reporting groups
Arm/Group | Acute Phase: Placebo TID | Acute Phase: Sodium Zirconium Cyclosilicate (ZS) 1.25 g TID | Acute Phase: ZS 2.5 g TID | Acute Phase: ZS 5 g TID | Acute Phase: ZS 10 TID | Total
Number analyzed (Participants) | 158 | 154 | 141 | 157 | 143 | 753
Age, Customized [Mean (Standard Deviation); unit: Years]
  Acute Phase | 65.6 (12.24) | 65.4 (13.07) | 65.9 (11.73) | 65.2 (11.91) | 66.2 (12.16) | 65.6 (12.24)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex/Gender, Customized. Gender by Acute Phase
  Participants
    Female | 60 | 71 | 50 | 61 | 63 | 305
    Male | 98 | 83 | 91 | 96 | 80 | 448
Race/Ethnicity, Customized [Number; unit: Participants] — Race/Ethnicity, Customized. Categories are not mutually exclusive
  Participants
    White | 136 | 131 | 125 | 132 | 120 | 644
    Black or African American | 17 | 20 | 11 | 20 | 19 | 87
    Asian | 2 | 0 | 5 | 3 | 2 | 12
    American Indian or Alaska Native | 2 | 0 | 0 | 1 | 1 | 4
    Native Hawaiian or other Pacific Islander | 1 | 3 | 0 | 0 | 1 | 5
    Other | 0 | 0 | 1 | 1 | 0 | 2
    Multiple Races | 0 | 0 | 1 | 0 | 0 | 1
Acute S-K baseline [Count of Participants; unit: Participants]
  ≤ 5.3 mmol/L | 95 | 76 | 72 | 90 | 94 | 427
  5.4-5.5 mmol/L | 22 | 38 | 29 | 36 | 27 | 152
  > 5.5 mmol/L | 41 | 40 | 40 | 31 | 22 | 174
Etiology of elevated S-K [Count of Participants; unit: Participants] — Etiology of elevated S-K. Categories are not mutually exclusive
  Participants
    Chronic kidney disease | 96 | 102 | 89 | 93 | 83 | 463
    Congestive heart failure | 66 | 57 | 54 | 64 | 59 | 300
    Diabetes mellitus | 96 | 94 | 84 | 96 | 81 | 451
    RAAS inhibitor medication | 101 | 109 | 97 | 99 | 96 | 502
Baseline eGFR [Count of Participants; unit: Participants] — Acute phase baseline - estimated Glomerular filtration rate (eGFR) Population: Subjects with non-missing acute phase baseline eGFR
  Participants
    <15 ml/min: number analyzed (Participants) | 158 | 151 | 138 | 154 | 143 | 744
    <15 ml/min | 15 | 8 | 15 | 8 | 10 | 56
    15-29+ ml/min: number analyzed (Participants) | 158 | 151 | 138 | 154 | 143 | 744
    15-29+ ml/min | 44 | 42 | 38 | 43 | 42 | 209
    30-59+ mL/min: number analyzed (Participants) | 158 | 151 | 138 | 154 | 143 | 744
    30-59+ mL/min | 61 | 73 | 48 | 64 | 50 | 296
    ≥60 mL/min: number analyzed (Participants) | 158 | 151 | 138 | 154 | 143 | 744
    ≥60 mL/min | 38 | 28 | 37 | 39 | 41 | 183

OUTCOME MEASURES:

1. Primary Outcome: Exponential Rate of Change in Serum Potassium (S-K) Levels During the Initial 48 Hours of Study Drug Treatment.
Time Frame: Through 48 hours acute phase
Population: ITT Population
Measure: Mean (Standard Error); unit: log(mmol/L)/hour
Groups:
- Acute Phase: ZS 10 g TID: Participants administered ZS 10 g TID as suspension orally for first 48 hours.
Arm/Group | Acute Phase: Placebo TID | Acute Phase: Sodium Zirconium Cyclosilicate (ZS) 1.25 g TID | Acute Phase: ZS 2.5 g TID | Acute Phase: ZS 5 g TID | Acute Phase: ZS 10 g TID
Number analyzed (Participants) | 158 | 154 | 141 | 157 | 143
log(mmol/L)/hour
  Through 24 Hours | -0.00128 (0.000243) | -0.00187 (0.000250) | -0.00205 (0.000263) | -0.00280 (0.000250) | -0.00382 (0.000258)
  Through 48 Hours | -0.00097 (0.000137) | -0.00110 (0.000141) | -0.00163 (0.000148) | -0.00223 (0.000141) | -0.00321 (0.000145)

2. Primary Outcome: Exponential Rate of Change in S-K Levels in the Subacute Phase.
Time Frame: Through 12 days subacute phase (Day 3 through Day 15)
Population: ITT population. One subject in the ZS 5 g TID/5 g QD group died on Study Day 4 and was excluded from the ITT Population
Measure: Mean (Standard Error); unit: log(mmol/L)/hour
Groups:
- Subacute Phase: Placebo Matched to ZS 1.25 g QD: Participants who received ZS 1.25 g TID in the acute phase and received placebo matched to ZS 1.25 g QD for 12 days.
- Subacute Phase: ZS 2.5 g ( Acute Phase: Placebo): Participants who received placebo in the acute phase and administered ZS 2.5 g as suspension QD for 12 days.
Arm/Group | Subacute Phase: Placebo Matched to ZS 1.25 g QD | Subacute Phase: ZS 1.25 g QD | Subacute Phase: Placebo Matched to ZS 2.5 g QD | Subacute Phase: ZS 2.5 g QD | Subacute Phase: Placebo Matched to ZS 5 g QD | Subacute Phase: ZS 5 g QD | Subacute Phase: Placebo Matched to ZS 10 g QD | Subacute Phase: ZS 10 g QD | Subacute Phase: ZS 1.25 (Acute Phase: Placebo) | Subacute Phase: ZS 2.5 g ( Acute Phase: Placebo)
Number analyzed (Participants) | 41 | 49 | 46 | 54 | 68 | 64 | 61 | 63 | 46 | 50
log(mmol/L)/hour
  Through Day 8 | 0.00054 (0.004803) | 0.00874 (0.004308) | 0.01104 (0.004123) | 0.00734 (0.003642) | 0.01441 (0.003776) | 0.00581 (0.003918) | 0.02469 (0.003939) | -0.00053 (0.003877) | 0.00643 (0.004171) | 0.00390 (0.004023)
  Through Day 15 | 0.00085 (0.001089) | 0.00198 (0.000959) | 0.00206 (0.001189) | 0.00237 (0.001049) | 0.00457 (0.001007) | 0.00089 (0.001049) | 0.00979 (0.001115) | 0.00136 (0.001097) | -0.00098 (0.001054) | 0.00023 (0.001004)

3. Secondary Outcome: Percentage of Subjects Who Achieve Normalization in S-K Levels After 48 Hours of Treatment
Time Frame: Through 48 hours acute phase
Population: Subjects from ITT population who have completed Acute phase
Measure: Number; unit: percentage of participants
Arm/Group | Acute Phase: Placebo TID | Acute Phase: Sodium Zirconium Cyclosilicate (ZS) 1.25 g TID | Acute Phase: ZS 2.5 g TID | Acute Phase: ZS 5 g TID | Acute Phase: ZS 10 g TID
Number analyzed (Participants) | 157 | 150 | 137 | 152 | 140
percentage of participants | 47.8 | 51.3 | 67.9 | 77.6 | 86.4

4. Secondary Outcome: Mean Change From Baseline in S-K at All Time Points Acute Phase
Description: Mean change from baseline in S-K at all time points over initial 48 hours
Time Frame: Through 48 hours acute phase. In particular, at Baseline; 1, 2, 4 hour Post 1st Dose on Study Day 1; 0 hour Pre-dose, 1, 4 hour Post 1st Dose on Study Day 2; and 0 hour Pre-dose on Study Day 3.
Population: ITT population
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Acute Phase: Placebo TID | Acute Phase: Sodium Zirconium Cyclosilicate (ZS) 1.25 g TID | Acute Phase: ZS 2.5 g TID | Acute Phase: ZS 5 g TID | Acute Phase: ZS 10 g TID
Number analyzed (Participants) | 158 | 154 | 141 | 157 | 143
mmol/L
  Baseline, mean | 5.30 (0.365) | 5.37 (0.369) | 5.35 (0.400) | 5.31 (0.337) | 5.26 (0.337)
  Study Day 1: 1 hour Post 1st Dose | 0.01 (0.404) | -0.01 (0.360) | -0.08 (0.394) | -0.06 (0.413) | -0.11 (0.361)
  Study Day 1: 2 hour Post 1st Dose | 0.00 (0.423) | -0.04 (0.366) | -0.06 (0.499) | -0.09 (0.355) | -0.18 (0.360)
  Study Day 1: 4 hour Post 1st Dose | -0.22 (0.429) | -0.28 (0.425) | -0.34 (0.409) | -0.31 (0.389) | -0.37 (0.445)
  Study Day 2: 0 hour Pre-dose | -0.18 (0.363) | -0.28 (0.393) | -0.32 (0.390) | -0.40 (0.375) | -0.52 (0.364)
  Study Day 2: 1 hour Post 1st Dose | -0.24 (0.484) | -0.27 (0.415) | -0.38 (0.479) | -0.46 (0.440) | -0.68 (0.437)
  Study Day 2: 4 hour Post 1st Dose | -0.22 (0.440) | -0.32 (0.449) | -0.40 (0.462) | -0.47 (0.465) | -0.62 (0.420)
  Study Day 3: 0 hour Pre-dose | -0.25 (0.413) | -0.30 (0.404) | -0.46 (0.398) | -0.54 (0.459) | -0.73 (0.496)

5. Secondary Outcome: Mean Percent Change From Baseline in S-K Change at All Time Points Acute Phase
Description: Mean percent change from baseline in S-K at all time points over initial 48 hours
Time Frame: Through 48 hours acute phase. In particular, 1, 2, 4 hour Post 1st Dose on Study Day 1; 0 hour Pre-dose, 1, 4 hour Post 1st Dose on Study Day 2; and 0 hour Pre-dose on Study Day 3.
Population: ITT population
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Acute Phase: Placebo TID | Acute Phase: Sodium Zirconium Cyclosilicate (ZS) 1.25 g TID | Acute Phase: ZS 2.5 g TID | Acute Phase: ZS 5 g TID | Acute Phase: ZS 10 g TID
Number analyzed (Participants) | 158 | 154 | 141 | 157 | 143
percentage
  Study Day 1: 1 hour Post 1st Dose Percent change | 0.09 (7.606) | -0.23 (6.732) | -1.37 (7.273) | -1.13 (7.791) | -2.08 (6.873)
  Study Day 1: 2 hour Post 1st Dose Percent change | 0.03 (7.911) | -0.81 (6.813) | -0.99 (9.384) | -1.71 (6.725) | -3.43 (6.779)
  Study Day 1: 4 hour Post 1st Dose Percent change | -4.05 (8.021) | -5.20 (7.842) | -6.34 (7.460) | -5.74 (7.283) | -6.91 (8.249)
  Study Day 2: 0 hour Pre-dose Percent change | -3.40 (6.819) | -5.14 (7.190) | -6.02 (7.099) | -7.31 (6.942) | -9.85 (6.693)
  Study Day 2: 1 hour Post 1st Dose Percent change | -4.42 (8.904) | -4.99 (7.717) | -6.95 (8.910) | -8.62 (8.082) | -12.70 (8.091)
  Study Day 2: 4 hour Post 1st Dose Percent change | -4.08 (8.253) | -5.82 (8.187) | -7.27 (8.405) | -8.63 (8.541) | -11.58 (7.645)
  Study Day 3: 0 hour Pre-dose Percent change | -4.62 (7.751) | -5.44 (7.476) | -8.48 (7.291) | -10.04 (8.33) | -13.76 (9.044)

6. Secondary Outcome: Time Subjects Remain Normokalemic (Subacute Phase)
Description: Time (number of days) subjects remain normokalemic (3.5 - 5.0 mmol/l) subacute phase
Time Frame: Through 18 days (12 days treatment, 6 days follow-up) of subacute phase
Population: ITT population. One subject (087-025) in the ZS 5 g TID/5 g QD group died on Study Day 4 and was excluded from the ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Subacute Phase: Placebo Matched to ZS 1.25 g QD | Subacute Phase: ZS 1.25 g QD | Subacute Phase: Placebo Matched to ZS 2.5 g QD | Subacute Phase: ZS 2.5 g QD | Subacute Phase: Placebo Matched to ZS 5 g QD | Subacute Phase: ZS 5 g QD | Subacute Phase: Placebo Matched to ZS 10 g QD | Subacute Phase: ZS 10 g QD | Subacute Phase: ZS 1.25 (Acute Phase: Placebo) | Subacute Phase: ZS 2.5 g (Acute Phase: Placebo)
Number analyzed (Participants) | 41 | 49 | 46 | 54 | 68 | 64 | 61 | 63 | 46 | 50
Days | 7.6 (4.71) | 7.2 (5.08) | 6.2 (4.78) | 8.6 (4.55) | 6.0 (4.43) | 9.0 (4.22) | 8.2 (4.64) | 10.2 (3.96) | 8.5 (4.57) | 8.2 (4.72)

7. Secondary Outcome: Percentage of Subjects Within Each Treatment Group Who Retained Normal S-K Values at End of Subacute Phase
Description: Percentage of subjects within each treatment group who retained normal S-K values (values between 3.5-5.0 mmol/L) at end of subacute phase
Time Frame: Through 18 days of subacute phase (12 days treatment, 6 days follow-up)
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Subacute Phase: Placebo Matched to ZS 1.25 g QD | Subacute Phase: ZS 1.25 g QD | Subacute Phase: Placebo Matched to ZS 2.5 g QD | Subacute Phase: ZS 2.5 g QD | Subacute Phase: Placebo Matched to ZS 5 g QD | Subacute Phase: ZS 5 g QD | Subacute Phase: Placebo Matched to ZS 10 g QD | Subacute Phase: ZS 10 g QD | Subacute Phase: ZS 1.25 (Acute Phase: Placebo) | Subacute Phase: ZS 2.5 g (Acute Phase: Placebo)
Number analyzed (Participants) | 41 | 49 | 46 | 54 | 68 | 64 | 61 | 63 | 46 | 50
percentage of participants | 73.2 | 59.2 | 65.2 | 64.8 | 54.4 | 57.8 | 60.7 | 61.9 | 67.4 | 66

8. Secondary Outcome: Mean Change From Subacute Baseline in Serum Potassium at All Time Points.
Description: Mean change from subacute baseline in serum potassium at all time points during subacute phase
Time Frame: Through 18 days of subacute phase (12 days treatment, 6 days follow-up)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Subacute Phase: Placebo Matched to ZS 1.25 g QD | Subacute Phase: ZS 1.25 g QD | Subacute Phase: Placebo Matched to ZS 2.5 g QD | Subacute Phase: ZS 2.5 g QD | Subacute Phase: Placebo Matched to ZS 5 g QD | Subacute Phase: ZS 5 g QD | Subacute Phase: Placebo Matched to ZS 10 g QD | Subacute Phase: ZS 10 g QD | Subacute Phase: ZS 1.25 (Acute Phase: Placebo) | Subacute Phase: ZS 2.5 g (Acute Phase: Placebo)
Number analyzed (Participants) | 41 | 49 | 46 | 54 | 68 | 64 | 61 | 63 | 46 | 50
mmol/L
  Acute Baseline, mean | 5.22 (0.263) | 5.29 (0.343) | 5.25 (0.268) | 5.23 (0.354) | 5.31 (0.302) | 5.24 (0.325) | 5.24 (0.290) | 5.27 (0.369) | 5.15 (0.293) | 5.19 (0.325)
  Subacute Baseline, mean | 4.81 (0.324) | 4.80 (0.391) | 4.77 (0.349) | 4.66 (0.336) | 4.76 (0.440) | 4.63 (0.357) | 4.42 (0.353) | 4.52 (0.448) | 4.81 (0.348) | 4.80 (0.379)
  Subacute Day 1 | 0.02 (0.362) | 0.15 (0.416) | 0.21 (0.416) | 0.11 (0.329) | 0.07 (0.493) | 0.12 (0.446) | 0.13 (0.363) | 0.00 (0.452) | 0.05 (0.373) | 0.04 (0.362)
  Subacute Day 2 | -0.06 (0.575) | 0.13 (0.405) | 0.07 (0.451) | 0.05 (0.360) | 0.12 (0.477) | 0.10 (0.519) | 0.28 (0.387) | 0.00 (0.531) | 0.07 (0.437) | 0.12 (0.389)
  Subacute Day 3 | 0.04 (0.387) | 0.11 (0.432) | 0.17 (0.431) | 0.18 (0.350) | 0.17 (0.503) | 0.11 (0.499) | 0.37 (0.426) | -0.06 (0.557) | 0.11 (0.400) | 0.03 (0.501)
  Subacute Day 6 | 0.11 (0.385) | 0.07 (0.411) | 0.22 (0.532) | 0.12 (0.356) | 0.27 (0.560) | 0.11 (0.510) | 0.43 (0.467) | 0.10 (0.573) | 0.04 (0.409) | 0.13 (0.457)
  Subacute Day 12 | 0.04 (0.477) | 0.18 (0.368) | 0.18 (0.520) | 0.23 (0.451) | 0.24 (0.584) | 0.14 (0.532) | 0.58 (0.485) | 0.06 (0.564) | -0.01 (0.438) | 0.04 (0.451)
  Subacute Day 18 | 0.06 (0.474) | 0.22 (0.459) | 0.09 (0.442) | 0.18 (0.522) | 0.26 (0.555) | 0.30 (0.539) | 0.59 (0.504) | 0.44 (0.652) | 0.09 (0.477) | 0.14 (0.492)

9. Secondary Outcome: Mean Percent Change From Subacute Baseline in Serum Potassium at All Time Points.
Description: Mean percent change from subacute baseline in serum potassium at all time points during subacute phase
Time Frame: Through 18 days of subacute phase (12 days treatment, 6 days follow-up)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Subacute Phase: Placebo Matched to ZS 1.25 g QD | Subacute Phase: ZS 1.25 g QD | Subacute Phase: Placebo Matched to ZS 2.5 g QD | Subacute Phase: ZS 2.5 g QD | Subacute Phase: Placebo Matched to ZS 5 g QD | Subacute Phase: ZS 5 g QD | Subacute Phase: Placebo Matched to ZS 10 g QD | Subacute Phase: ZS 10 g QD | Subacute Phase: ZS 1.25 (Acute Phase: Placebo) | Subacute Phase: ZS 2.5 g (Acute Phase: Placebo)
Number analyzed (Participants) | 41 | 49 | 46 | 54 | 68 | 64 | 61 | 63 | 46 | 50
percentage
  Subacute Day 1 Percent Change | 0.66 (7.386) | 3.31 (8.848) | 4.74 (8.819) | 2.58 (7.055) | 2.03 (9.511) | 2.90 (9.738) | 3.15 (8.368) | 0.45 (9.412) | 1.26 (7.859) | 0.99 (7.696)
  Subacute Day 2 Percent Change | -1.05 (12.031) | 2.79 (8.465) | 1.79 (9.198) | 1.30 (7.766) | 2.96 (8.913) | 2.54 (11.925) | 6.58 (8.908) | 0.67 (11.555) | 1.59 (8.948) | 2.67 (8.257)
  Subacute Day 3 Percent Change | 1.15 (7.930) | 2.56 (9.098) | 3.79 (8.956) | 4.12 (7.870) | 4.15 (9.464) | 2.82 (11.259) | 8.73 (9.982) | -0.52 (11.590) | 2.49 (8.510) | 1.12 (10.533)
  Subacute Day 6 Percent Change | 2.46 (8.048) | 1.58 (8.271) | 4.83 (10.881) | 2.90 (7.769) | 6.16 (11.061) | 2.84 (11.565) | 10.22 (11.027) | 2.90 (12.396) | 1.18 (8.583) | 3.05 (9.397)
  Subacute Day 12 Percent Change | 1.13 (9.955) | 3.95 (7.550) | 4.16 (10.727) | 5.33 (9.976) | 5.67 (12.400) | 3.53 (11.664) | 13.52 (11.493) | 1.88 (12.344) | 0.07 (9.117) | 1.10 (9.679)
  Subacute Day 18 Percent Change | 1.56 (10.145) | 4.73 (10.015) | 2.19 (9.338) | 4.35 (11.587) | 6.00 (11.393) | 7.07 (11.918) | 13.80 (12.182) | 10.38 (14.581) | 1.94 (10.241) | 3.01 (10.301)

ADVERSE EVENTS:
Time Frame: Seven days after the last dose of study medication. 21 days overall
Groups:
- Subacute Phase: ZS 1.25 g QD (Acute Phase: Placebo): Participants who received placebo in the acute phase and administered ZS 1.25 g as suspension QD for 12 days.
- Subacute Phase: ZS 2.5 g QD (Acute Phase; Placebo): Participants who received placebo in the acute phase and administered ZS 2.5 g as suspension QD for 12 days.
Arm/Group | Acute Phase: Placebo TID | Acute Phase: Sodium Zirconium Cyclosilicate (ZS) 1.25 g TID | Acute Phase: ZS 2.5 g TID | Acute Phase: ZS 5 g TID | Acute Phase: ZS 10 TID | Subacute Phase: Placebo Matched to ZS 1.25g QD | Subacute Phase: ZS 1.25 g QD | Subacute Phase: Placebo Matched to ZS 2.5 g QD | Subacute Phase: ZS 2.5 g QD | Subacute Phase: Placebo Matched to ZS 5 g QD | Subacute Phase: ZS 5 g QD | Subacute Phase: Placebo Matched to ZS 10 g QD | Subacute Phase: ZS 10 g QD | Subacute Phase: ZS 1.25 g QD (Acute Phase: Placebo) | Subacute Phase: ZS 2.5 g QD (Acute Phase; Placebo)
Serious Adverse Events (participants affected / at risk) | 1/158 | 0/154 | 0/141 | 0/157 | 0/143 | 1/41 | 2/49 | 1/46 | 2/54 | 2/68 | 3/65 | 1/61 | 1/63 | 1/46 | 1/50
Other Adverse Events (participants affected / at risk) | 9/158 | 18/154 | 6/141 | 6/157 | 10/143 | 14/41 | 10/49 | 7/46 | 13/54 | 12/68 | 14/65 | 6/61 | 16/63 | 8/46 | 6/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Acute Phase: Placebo TID (N=158) | Acute Phase: Sodium Zirconium Cyclosilicate (ZS) 1.25 g TID (N=154) | Acute Phase: ZS 2.5 g TID (N=141) | Acute Phase: ZS 5 g TID (N=157) | Acute Phase: ZS 10 TID (N=143) | Subacute Phase: Placebo Matched to ZS 1.25g QD (N=41) | Subacute Phase: ZS 1.25 g QD (N=49) | Subacute Phase: Placebo Matched to ZS 2.5 g QD (N=46) | Subacute Phase: ZS 2.5 g QD (N=54) | Subacute Phase: Placebo Matched to ZS 5 g QD (N=68) | Subacute Phase: ZS 5 g QD (N=65) | Subacute Phase: Placebo Matched to ZS 10 g QD (N=61) | Subacute Phase: ZS 10 g QD (N=63) | Subacute Phase: ZS 1.25 g QD (Acute Phase: Placebo) (N=46) | Subacute Phase: ZS 2.5 g QD (Acute Phase; Placebo) (N=50)
Diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nocardiosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hospitalization (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Acute Phase: Placebo TID (N=158) | Acute Phase: Sodium Zirconium Cyclosilicate (ZS) 1.25 g TID (N=154) | Acute Phase: ZS 2.5 g TID (N=141) | Acute Phase: ZS 5 g TID (N=157) | Acute Phase: ZS 10 TID (N=143) | Subacute Phase: Placebo Matched to ZS 1.25g QD (N=41) | Subacute Phase: ZS 1.25 g QD (N=49) | Subacute Phase: Placebo Matched to ZS 2.5 g QD (N=46) | Subacute Phase: ZS 2.5 g QD (N=54) | Subacute Phase: Placebo Matched to ZS 5 g QD (N=68) | Subacute Phase: ZS 5 g QD (N=65) | Subacute Phase: Placebo Matched to ZS 10 g QD (N=61) | Subacute Phase: ZS 10 g QD (N=63) | Subacute Phase: ZS 1.25 g QD (Acute Phase: Placebo) (N=46) | Subacute Phase: ZS 2.5 g QD (Acute Phase; Placebo) (N=50)
Atrial fibrilliation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 5 | 2 | 3 | 1 | 0 | 0 | 2 | 2 | 3 | 2 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 5 | 0 | 1 | 0 | 4 | 4 | 1 | 3 | 0 | 5 | 0 | 4 | 3 | 0
Urinary tract infection, bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
ZS Pharma has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.